CLINICAL TRIAL: NCT06460792
Title: The Quality of Ultrasound-guided Peripheral Nerve Blocks, Nerve Injury, Bleeding Complications and Learning - a Prospective Observational Cohort Study
Brief Title: Ultrasound-guided Peripheral Nerve Blocks - a Database
Acronym: Blockbase
Status: Recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: p-2024-15805
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Regional Anesthesia
Keywords: nerve block; ultrasound guidance; complications; nerve injury; bleeding; success rate; learning
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound-guided peripheral nerve block — Ultrasound-guided peripheral nerve blocks. Registration of quality, complications and learning as detailed in the description

SUMMARY:
Peripheral nerve blocks are often used in anaesthesia. They can be used as the only method of anaesthesia during surgery or in combination with other methods, e.g., general anaesthesia and sedation. Moreover, peripheral nerve blocks are used to treat postoperative pain, alleviate pain in trauma patients, and for painful procedures.

For a method to be clinically useful, it is essential to understand the factors contributing to high success rates. It is equally important to know the complications related to the method. Finally, it is essential to establish a robust learning system where the anesthesiologists can track their nerve block performance over time and compare it to high performers and general performance. Therefore, we aim to establish a prospective and ongoing database to gain insight into 1) Factors contributing to block quality, e.g., success rate and nerve block duration; 2) Frequencies and types of nerve injuries and bleeding complications associated with the block procedure; 3) Tracking of block performance by anaesthesiologists.

DETAILED DESCRIPTION:
Introduction Peripheral nerve blocks are often used in anaesthesia. They can be used as the only method of anaesthesia during surgery or in combination with other methods, e.g., general anaesthesia and sedation. Moreover, peripheral nerve blocks are used to treat postoperative pain, alleviate pain in trauma patients, and for painful procedures.

For a method to be clinically useful, it is essential to understand the factors contributing to high success rates. It is equally important to know the complications related to the method. Finally, it is essential to establish a robust learning system where the anesthesiologists can track their nerve block performance over time and compare it to high performers and general performance. Therefore, we aim to establish a prospective and ongoing database to gain insight into 1) Factors contributing to block quality, e.g., success rate and nerve block duration; 2) Frequencies and types of nerve injuries and bleeding complications associated with the block procedure; 3) Tracking of block performance by anaesthesiologists. These three points are described in more detail below:

1. Success rate (block quality) It is difficult to get an overview of the success rates of peripheral nerve blocks. Most studies focus on one specific nerve block, and the number of included patients is often low. In addition, the block procedure is performed by a few anaesthesiologists who are highly skilled in the specific procedure. By establishing a database, including the most used peripheral nerve blocks used in different settings, i.e., surgery, perioperative pain management, and painful procedures, and by including anaesthesiologists with varying levels of experience and expertise, it will be possible to get a more detailed picture of factors that are important for achieving high success rates.
2. Complications Nerve injury. Peripheral nerve blocks are generally considered safe to use with low complication rates. However, complications can be severe and result in permanent nerve injury. Therefore, it is essential to get an overview of block-related complications and factors associated with these complications. Different regions have specific characteristics, and complications probably follow a characteristic pattern. A database with sufficient data will allow us to detail essential factors for understanding how complications develop and turn into permanent injuries.

   Bleeding. Today, many patients receive anticoagulant therapy. We will, therefore, collect data on bleeding complications associated with the block procedure.
3. Learning Ultrasound-guided peripheral nerve blocks require a certain amount of skill to deposit LA in the correct place. By gathering data on block quality from individual anaesthesiologists over time it will be possible to gain insight into learning curves and factors important for learning different block procedures.

Methods Study design: Observational prospective cohort study. Setting: Initially, a single-centre study at the Department of Anaesthesiology, North Zealand Hospital. We envision to include as many centres as possible in Denmark.

Participants: Patients scheduled for peripheral nerve blocks. Prior to collecting follow-up data, informed consent will be obtained from each participant through an automated and secure sms system.

Variables: The following variables are registered:

Patient demographics: Social security number, age, sex, height, weight, comorbidity (diabetes, use of insulin, chronic pain, pain medication, anticoagulant medication), ASA status, and type of surgery performed.

Technical block data: Date and time for the peripheral nerve block, performing anaesthesiologist, block details (name of block, type of LA, volume of LA, concentration of LA, anatomical location of LA injection, adjuvants used, onset time).

Peripheral nerve block quality and success rate: success rate, need of supplementary blocks, use of tourniquet, reasons for block deemed unsuccessful.

Bleeding complications: details on bleeding complications associated with the block procedure.

Follow-up by surveys:

Day 1: duration of peripheral nerve block, pain after block termination. Day 2: measures if block duration > 24 h. Day 30: signs of nerve injury: altered sensation, pain, decreased muscle force. Day 90: continuous signs of nerve injury: altered sensation, pain, decreased muscle force.

Day 365: continuous signs of nerve injury: altered sensation, pain, decreased muscle force.

Data sources/measurements: All variables are part of data that are normally registered for patients who have a peripheral nerve block. However, the purpose of establishing the database is to perform a systematic data capture. We will use the secure web application for online research databases, REDCap to enter data through electronic CRFs and through surveys sent to the patients (follow-up).

Study size: The purpose of establishing the database is to continuously register peripheral nerve blocks in patients. As such there is no pre-defined study size.

Statistical methods: We will use descriptive statistics and inferential statistical analyses, e.g., regression analyses, etc.

ELIGIBILITY:
Inclusion Criteria:

- age > 2 years

Exclusion Criteria

* Infection at puncture site
* Allergy to local anesthetics
* Unable to understand given oral instruction

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with a peripheral nerve block as part of their normal treatment
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2029-06-04 (Estimated); Study Completion 2029-06-04 (Estimated)

PRIMARY OUTCOMES:
Block Success | 2 hours
  Clinical evaluation of nerve function

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rothe, MD, Principal Investigator — Nordsjællands Hospital Hillerød
Locations (1):
- Dept of Anesthesiology, Nordsjællands Hospital, Hillerød, Denmark